CLINICAL TRIAL: NCT06442306
Title: Development of a Pain Neuroscience Education Program for Patients Who Are Opioid Dependence With Concurrent Chronic Musculoskeletal Pain
Brief Title: Evaluation of Pain Neuroscience Education for Patients Who Experience Chronic Pain With Concurrent Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wichita State University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Nicole D Windsor, Physical Therapist, PhD student, Teaching assistant, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53966
Record Dates: First submitted 2024-05-09; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Opioid Dependence
Keywords: Chronic Musculoskeletal Pain; Opioid Dependence; Pain Neuroscience Education; Neurophysiology of Pain Questionnaire; Pain Self-Efficacy Questionnaire; Tampa Scale for Kinesiophobia
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study with a Pain Neuroscience Education group and a General Health Education group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education group (Experimental): The PNE group received the a-PNE education curriculum which was created with patient-friendly verbiage and used to educate subjects about the inner workings of the nervous system. The a-PNE curriculum, a PowerPoint presentation was divided into four, 15-minute, one-on-one sessions with the PI in a private treatment room to facilitate discussion and minimize distractions. The educational information was related directly to the patients' CMP/OpD experience to personalize the intervention and presented at a pace that was appropriate for each patient. At the conclusion of each session, the PNE group was provided handouts containing information that was reviewed during that session. At the end of the a-PNE intervention, the patients completed the three questionnaires.
  Interventions: Other: Pain Neuroscience Education
- General Health Education group (Active Comparator): The GHE group was provided practical education for healthy living over four monthly sessions, 15-minutes per session. The GHE intervention was comprised of topics promoting healthy living in a one-on-one session with the PI in a private treatment room to facilitate discussion. At the conclusion of each session, the GHE group was provided handouts containing information that was reviewed during the session. At the end of the GHE intervention, the patients completed the three questionnaires.
  Interventions: Other: General Health Education

INTERVENTIONS:
Other: Pain Neuroscience Education — Pain Neuroscience Education (PNE) is a cognitive-based education intervention that aims to change pain beliefs in patients experiencing CMP. Researchers have found PNE beneficial in assisting patients to reframe their understanding, attitudes, thoughts, and beliefs regarding their pain experience. PNE directs patients to relate chronic pain to overly sensitive nerves rather than assumed tissue damage. Further, PNE encourages patients to perform daily activities, work, and function in society, all despite pain. This facilitates behavior changes that are key in amending a patient's biopsychosocial state. Multiple sources make a strong case for the incorporation of PNE in having positive effects on reducing physical disability and modulating fear and anxiety in patients with CMP. Researchers have established a positive influence of PNE toward decreased kinesiophobia and have demonstrated a relation between increased self-efficacy and increased functional ability.
  Other Names: Neuroscience Education; Biopsychosocial pain education; Pain neurophysiology education; Pain science education; Therapeutic neuroscience education
  Arms: Pain Neuroscience Education group
Other: General Health Education — General Health Education included: 20 Benefits of Walking 30 Minutes a Day; Why You Should Quit: Smoking Cessation; Heat vs. Cold: How to Use it For Pain Control; Sleep Hygiene.
  Arms: General Health Education group

SUMMARY:
Chronic musculoskeletal pain (CMP) is estimated to affect over 100 million adults and is targeted as an instigator of opioid dependence (OpD). Opioid medications are often the first response for patients suffering with CMP; yet over 10 million people admit to misusing opioids annually. With the opioid epidemic, the healthcare system now has a population of patients who experience CMP with concurrent OpD (CMP/OpD). This persistent problem can create a perfect storm of kinesiophobia, reduced self-efficacy, and physical dysfunction. A critical component to chronic pain management is understanding how patients view their pain experience. Education may be one key that unlocks the door to functional improvement, but traditional physical therapy (PT) education utilizes anatomical models that focus on tissue damage and peripheral sources of pain. Researchers have explored educating people about pain via Pain Neuroscience Education (PNE), a cognitive-based intervention that facilitates understanding of the biological processes underpinning the pain state. PNE may facilitate understanding pain experiences that are normal and expected, with the intent to reduce fear and increase pain self-efficacy. As yet, utilization of PNE has not been researched in patients with CMP/OpD. Therefore, authors hypothesize that the introduction of an adapted PNE (a-PNE) curriculum, as a single intervention, may facilitate positive changes in kinesiophobia, pain self-efficacy, and knowledge of the neurophysiology of pain for patients with CMP/OpD.

DETAILED DESCRIPTION:
Methods Study Design This study was a pre-test-post-test, quasi-experimental design with patients suffering from CMP/OpD being treated at a family practice clinic associated with University of Kentucky. A quasi-experimental study was chosen due to the small sample of convenience.

Patients Patients were recruited from an opioid management program (OMP) at the referenced family practice clinic. At the time of study recruitment, the OMP had 31 patients participating monthly.

Procedures The 21 participating patients were divided into two groups via a coin toss; 13 were included in the experimental group (PNE) and eight were included in the general health education control group (GHE).

All patients reviewed and signed the IRB approved consent/HIPAA form and performed the MMSE. Each patient completed the Tampa Scale of Kinesiophobia (TSK-11), Pain Self-Efficacy Questionnaire (PSEQ), and the Neurophysiology of Pain Questionnaire (NPQ) at the onset of the study. All intervention sessions were completed once per month directly after the patient's regularly scheduled monthly OMP appointment.

The PNE group received the a-PNE curriculum which was created with patient-friendly verbiage and used to educate subjects about the inner workings of the nervous system. The a-PNE curriculum, a PowerPoint presentation was divided into four, 15-minute, one-on-one sessions with the PI in a private treatment room to facilitate discussion and minimize distractions. The educational information was related directly to the patients' CMP/OpD experience to personalize the intervention and presented at a pace that was appropriate for each patient. At the conclusion of each session, the PNE group was provided handouts containing information that was reviewed during that session. At the end of the a-PNE intervention, the patients completed the three questionnaires.

The GHE group was provided practical education for healthy living over four monthly sessions, 15-minutes per session. The GHE intervention was comprised of topics promoting healthy living in a one-on-one session with the PI in a private treatment room to facilitate discussion. At the conclusion of each session, the GHE group was provided handouts containing information that was reviewed during the session. At the end of the GHE intervention, the patients completed the three questionnaires.

It should be noted that no patients were receiving other physical therapy interventions throughout the time of the study. The principal investigator removed exercise-related language and overt physical therapy-related topics to focus primarily on the psychosocial constructs for both groups. Considering the many factors surrounding this cohort, multiple sessions were chosen for the two groups to minimize the effects of CMP/OpD of decreased attention span, decreased working memory and decreased cognitive flexibility, which has been demonstrated in the literature.

Ninety days after the completion of the intervention sessions and the post-program assessments, a follow-up data collection was performed in which all patients completed the three questionnaires. After the research study was complete and all data collected, the GHE subjects were offered the identical a-PNE intervention which was utilized with the PNE group.

Statistical Analysis Statistical analyses were performed using the SPSS software (v.27.0, SPSS, Inc., Chicago, IL, USA). The significance level was set at P<0.05. The scores of three patients who did not complete the study were removed from the data set.

Normative distribution was evaluated utilizing the Shapiro-Wilk test. Descriptive statistics, including means and standard deviations (SD), were gathered for baseline demographic data. A group (a-PNE or GHE) by time (pre-intervention, post-intervention, and 90-day post-intervention) interaction analysis of variance (ANOVA) was completed for each dependent variable. Analysis included the Mauchly's Test of Sphericity to correct for violations. Bonferroni's correction was used as needed. Pearson's correlation was performed to inquire of correlation between variables.

Paired samples t-tests were conducted on each group and utilized to analyze pre-intervention to post-intervention and pre-intervention to 90-day post-intervention scores for each of the three dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were actively participating in an Opioid Management Program.

Exclusion Criteria:

* 18 years of age or younger
* Score of 24 or less on the Mini Mental State Examination

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Pre-intervention (baseline), post-intervention (4-months past baseline), and 90-day post-intervention (7-months past baseline)
  Kinesiophobia was measured by the 11-question TSK-11. Kinesiophobia is the fear of movement, or the fear of pain associated with movement. Subjects rate each item on a 4-point Likert scale with scoring ranging from "strongly disagree" to "strongly agree". The TSK-11 tool specifically assesses a subject's fear of pain due to movement and is a valid and reliable tool for measuring kinesiophobia. The highest score available on the TSK-11 is 44 points, with higher scores indicating increased fear. The minimum detectible change (MDC) for the TSK-11 is 5.6, minimal clinically important difference (MCID) is 6 points, and test-retest reliability is 0.81 (95% CI, 0.58-0.93).
Pain Self-Efficacy Questionnaire (PSEQ) | Pre-intervention (baseline), post-intervention (4-months past baseline), and 90-day post-intervention (7-months past baseline)
  The patient's confidence with function despite pain, or self-efficacy, was measured by the Pain Self-Efficacy Questionnaire (PSEQ). The PSEQ measures a patient's confidence in performing certain tasks, despite pain, and has a maximum score of 60 points which relates to the most positive outcome for the subject (with zero being the lowest self-efficacy). The PSEQ is a valid and reliable tool for measuring pain self-efficacy with a test-retest reliability of 0.85 (95% CI, 0.74-0.92), MDC of 10.9 and MCID of 11 points.
Neurophysiology of Pain Questionnaire | Pre-intervention (baseline), post-intervention (4-months past baseline), and 90-day post-intervention (7-months past baseline)
  Knowledge gained and retained regarding the neurophysiology supporting the CMP experience was measured via the Neurophysiology of Pain Questionnaire (NPQ). The NPQ is a 12-item assessment that seeks to measure how a subject understands the biological mechanisms that sustain the pain experience. Statements are answered true, false, or unsure. There are 12 points possible with a higher score indicating more retained pain knowledge. Post-intervention, the NPQ will ascertain the subject's understanding of the a-PNE curriculum. The NPQ currently has no test-retest reliability, MDC or MCID available.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Harrison, PhD, Study Chair — University of Kentucky; Nicole D Windsor, PhD, Principal Investigator — University of Kentucky; Tony English, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Inquiries can be made to principal investigator. Study protocol, Subject de-identified demographics, outcome measure scores, statistical analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data is available at any time.
Access Criteria: Data can be accessed by emailing nicole.windsor@wichita.edu

REFERENCES:
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Louw A, Puentedura EL, Mintken P. Use of an abbreviated neuroscience education approach in the treatment of chronic low back pain: a case report. Physiother Theory Pract. 2012 Jan;28(1):50-62. doi: 10.3109/09593985.2011.562602. Epub 2011 Jul 3. PMID 21721995
- [Background] Louw A, Zimney K, O'Hotto C, Hilton S. The clinical application of teaching people about pain. Physiother Theory Pract. 2016 Jul;32(5):385-95. doi: 10.1080/09593985.2016.1194652. Epub 2016 Jun 28. PMID 27351903
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Lluch E, Duenas L, Falla D, Baert I, Meeus M, Sanchez-Frutos J, Nijs J. Preoperative Pain Neuroscience Education Combined With Knee Joint Mobilization for Knee Osteoarthritis: A Randomized Controlled Trial. Clin J Pain. 2018 Jan;34(1):44-52. doi: 10.1097/AJP.0000000000000511. PMID 28514231
- [Background] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Fernandez-Carnero J, La Touche R. Manual Therapy, Therapeutic Patient Education, and Therapeutic Exercise, an Effective Multimodal Treatment of Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):887-97. doi: 10.1097/PHM.0000000000000293. PMID 25888653
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503
- [Background] Souza CM, Martins J, Libardoni TC, de Oliveira AS. Self-efficacy in patients with chronic musculoskeletal conditions discharged from physical therapy service: A cross-sectional study. Musculoskeletal Care. 2020 Sep;18(3):365-371. doi: 10.1002/msc.1469. Epub 2020 Apr 8. PMID 32267617
- [Background] Tsuji H, Tetsunaga T, Tetsunaga T, Nishida K, Misawa H, Ozaki T. The factors driving self-efficacy in intractable chronic pain patients: a retrospective study. J Orthop Surg Res. 2019 Dec 30;14(1):473. doi: 10.1186/s13018-019-1535-9. PMID 31888662
- [Background] Archer KR, Phelps KD, Seebach CL, Song Y, Riley LH 3rd, Wegener ST. Comparative study of short forms of the Tampa Scale for Kinesiophobia: fear of movement in a surgical spine population. Arch Phys Med Rehabil. 2012 Aug;93(8):1460-2. doi: 10.1016/j.apmr.2012.03.024. Epub 2012 Apr 3. PMID 22481127
- [Background] Mintken PE, Cleland JA, Whitman JM, George SZ. Psychometric properties of the Fear-Avoidance Beliefs Questionnaire and Tampa Scale of Kinesiophobia in patients with shoulder pain. Arch Phys Med Rehabil. 2010 Jul;91(7):1128-36. doi: 10.1016/j.apmr.2010.04.009. PMID 20599053
- [Background] Hapidou EG, O'Brien MA, Pierrynowski MR, de Las Heras E, Patel M, Patla T. Fear and Avoidance of Movement in People with Chronic Pain: Psychometric Properties of the 11-Item Tampa Scale for Kinesiophobia (TSK-11). Physiother Can. 2012 Summer;64(3):235-41. doi: 10.3138/ptc.2011-10. PMID 23729957
- [Background] Briet JP, Bot AG, Hageman MG, Menendez ME, Mudgal CS, Ring DC. The pain self-efficacy questionnaire: validation of an abbreviated two-item questionnaire. Psychosomatics. 2014 Nov-Dec;55(6):578-85. doi: 10.1016/j.psym.2014.02.011. Epub 2014 Feb 28. PMID 25016359
- [Background] Chiarotto A, Falla D, Polli A, Monticone M. Validity and Responsiveness of the Pain Self-Efficacy Questionnaire in Patients With Neck Pain Disorders. J Orthop Sports Phys Ther. 2018 Mar;48(3):204-216. doi: 10.2519/jospt.2018.7605. Epub 2017 Dec 19. PMID 29257925
- [Background] Chiarotto A, Vanti C, Cedraschi C, Ferrari S, de Lima E Sa Resende F, Ostelo RW, Pillastrini P. Responsiveness and Minimal Important Change of the Pain Self-Efficacy Questionnaire and Short Forms in Patients With Chronic Low Back Pain. J Pain. 2016 Jun;17(6):707-18. doi: 10.1016/j.jpain.2016.02.012. Epub 2016 Mar 11. PMID 26975193
- [Background] Catley MJ, O'Connell NE, Moseley GL. How good is the neurophysiology of pain questionnaire? A Rasch analysis of psychometric properties. J Pain. 2013 Aug;14(8):818-27. doi: 10.1016/j.jpain.2013.02.008. Epub 2013 May 4. PMID 23651882
- [Background] Vaughan B, Mulcahy J, Fitzgerald K, Austin P. Evaluating Patient's Understanding of Pain Neurophysiology: Rasch Analysis of the Neurophysiology of Pain Questionnaire. Clin J Pain. 2019 Feb;35(2):133-139. doi: 10.1097/AJP.0000000000000658. PMID 30260841
- [Background] van Ittersum MW, van Wilgen CP, van der Schans CP, Lambrecht L, Groothoff JW, Nijs J. Written pain neuroscience education in fibromyalgia: a multicenter randomized controlled trial. Pain Pract. 2014 Nov;14(8):689-700. doi: 10.1111/papr.12137. Epub 2013 Nov 20. PMID 24251724
- [Background] Wijma AJ, Speksnijder CM, Crom-Ottens AF, Knulst-Verlaan JMC, Keizer D, Nijs J, van Wilgen CP. What is important in transdisciplinary pain neuroscience education? A qualitative study. Disabil Rehabil. 2018 Sep;40(18):2181-2191. doi: 10.1080/09638288.2017.1327990. Epub 2017 May 19. PMID 28524700
- [Background] Tellez-Garcia M, de-la-Llave-Rincon AI, Salom-Moreno J, Palacios-Cena M, Ortega-Santiago R, Fernandez-de-Las-Penas C. Neuroscience education in addition to trigger point dry needling for the management of patients with mechanical chronic low back pain: A preliminary clinical trial. J Bodyw Mov Ther. 2015 Jul;19(3):464-72. doi: 10.1016/j.jbmt.2014.11.012. Epub 2014 Nov 22. PMID 26118519
- [Background] Amer-Cuenca JJ, Pecos-Martin D, Martinez-Merinero P, Lluch Girbes E, Nijs J, Meeus M, Ferrer Pena R, Fernandez-Carnero J. How Much Is Needed? Comparison of the Effectiveness of Different Pain Education Dosages in Patients with Fibromyalgia. Pain Med. 2020 Apr 1;21(4):782-793. doi: 10.1093/pm/pnz069. PMID 31216027
- [Background] Louw A, Puentedura EJ, Zimney K, Schmidt S. Know Pain, Know Gain? A Perspective on Pain Neuroscience Education in Physical Therapy. J Orthop Sports Phys Ther. 2016 Mar;46(3):131-4. doi: 10.2519/jospt.2016.0602. PMID 26928735
- [Background] Louw A, Sluka KA, Nijs J, Courtney CA, Zimney K. Revisiting the Provision of Pain Neuroscience Education: An Adjunct Intervention for Patients but a Primary Focus of Clinician Education. J Orthop Sports Phys Ther. 2021 Feb;51(2):57-59. doi: 10.2519/jospt.2021.9804. Epub 2020 Oct 19. PMID 33076759

DOCUMENTS (1):
  • Informed Consent Form (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT06442306/ICF_000.pdf